CLINICAL TRIAL: NCT06105684
Title: Phase II Single Arm Trial of Low Dose Capecitabine in Patients With Advanced Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Humaria Sarfraz, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300012026 (UAB23115); Robert Award (Other: UAB Cancer Center); Breast Cancer Foundation (Other: Breast Cancer Foundation)
Record Dates: First submitted 2023-10-23; First posted 2023-10-30 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Low dose capecitabine (Xeloda) (Experimental): 1000 mg capecitabine daily by mouth.
  Interventions: Drug: Capecitabine Pill

INTERVENTIONS:
Drug: Capecitabine Pill — Will be given once per day by mouth
  Other Names: Xeloda

SUMMARY:
This is a phase II study aiming at evaluating capecitabine prospectively at a dose of 1000 mg once daily in patients with advanced breast cancer who are ≥60 years of age, or frail at any age, with a greater risk of complications and poorer outcomes with other treatments.

DETAILED DESCRIPTION:
The study is a phase II, single arm study in which all patients will receive the study drug. Participants will include older/frail patients with metastatic breast cancer.

All patients will be treated with capecitabine 1000 mg daily. There will be a total of 40 participants with measurable disease on this trial.

The study will encompass participants with locally advanced unresectable/metastatic breast cancer with measurable disease, who progressed on at least 1 prior therapy in the metastatic setting. Breast cancer subtypes include HR+ HER2 negative, or TNBC, age ≥ 60 years old, or frail patients at a younger age. ECOG PS 0- 2.

The study will discontinue if progressive disease or unacceptable toxicity is noted.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed breast cancer with HER2 negative status. A copy of the pathology report is required at the time of enrollment.

   1. HER2 negativity will be determined by in situ hybridization (ISH) non- amplified and IHC 0 or 1+ or 2+.
   2. Patients with HR (hormone receptor) positive and triple negative breast cancer (TNBC) will be eligible for enrollment.
2. Metastatic or locally advanced breast cancer, with at least one measurable lesion according to RECIST (v1.1).
3. ECOG performance status of 0-2.
4. Patients must have progressed on at least 1 prior line of therapy in the metastatic setting (hormonal therapy or chemotherapy)
5. Adequate organ function as evidenced by:

   1. ANC >1.5 x 10⁹/L (1500/µL) or > 1.3 x 10⁹/L (1300/µL) for patients with history of benign ethnic neutropenia.
   2. Platelet count ≥100,000/µL (without transfusion within 2 weeks prior to initiation of study treatment (Cycle 1, day 1)).
   3. Hemoglobin ≥9.0 g/dl. Patients may be transfused or receive erythropoietic treatment to meet this criterion.
   4. AST, ALT, and alkaline phosphatase ≤2.5 x upper limit of normal (ULN) with following exceptions: I. Patients with documented liver metastasis: AST and ALT ≤5 x ULN II. Patients with documented liver or bone metastasis: alkaline phosphatase ≤5 x ULN
   5. Serum bilirubin ≤1.5 x ULN

      • Patients with known Gilbert disease who have serum bilirubin level ≤3 x ULN may be enrolled.
   6. INR and aPTT ≤1.5 x ULN

      • This applies only to the patients who are not receiving therapeutic anticoagulation; patients receiving therapeutic anticoagulation should be on a stable dose.
   7. Creatinine clearance > 30 mL/min (measured using Cockcroft-Gault equation or estimated glomerular filtration rate from the Modification of Diet in Renal Disease Study)
6. Patients must be able to provide signed informed consent.
7. Female patients of any ethnic group. Female patients must be surgically sterile, postmenopausal (no menses for at least one year), or using medically approved method of contraception (excluding rhythm, withdraw or abstinence). Men must agree to use a medically approved method of contraception (excluding rhythm, withdraw or abstinence).
8. Patients ≥60 years old and/or frail patients at any age, defined by the investigator as an individual at greater risk of complications and poorer outcomes with systemic therapy, secondary to a lower physiologic reserve and higher comorbidities and functional deficits.
9. Complete initial work-up within 2 weeks prior to start of treatment (Cycle 1 Day 1).
10. Patients known to be HIV positive are eligible if they meet the inclusion criteria.

Exclusion Criteria:

1. Any history of treatment with Capecitabine in metastatic setting.
2. Patients who only have non-measurable disease.
3. Patients with severe hepatic (bilirubin > 3 times upper limit of normal) or renal failure (CrCl < 30 calculated using Cockcroft-Gault formula).
4. Patients who are unable to swallow pills
5. Patients with HER2 positive breast cancer
6. Major surgical procedure within 3 weeks prior to study entry.
7. Spinal cord compression not definitively treated with surgery and/or radiation, or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for >2 weeks prior to initiation of study treatment (Cycle 1, Day 1)

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (RR) evaluation | Baseline up to 12 weeks
  Evaluate response rate (RR) as defined per Response Evaluation Criteria in Solid Tumors (RECIST) criteria (v 1.1). Response and progression of disease will be evaluated in this study using the international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee; version 1.1. Patients will be evaluated for response every 12 weeks per RECIST Criteria.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 36 months
  Initiation of treatment to the occurrence of disease progression or death. The RECIST v. 1.1 criteria will be used to evaluate progression-free survival as well as CT and PET scans. Baseline to the date of first documented progression to date of death from any cause, whichever comes first, assessed up to 36 months.
Overall survival (OS) | Baseline up to 36 months
  The time which begins at diagnosis (or at the start of treatment) and up to the time of death.
Number of adverse events | Baseline up to 36 months
  Incidence of Treatment-Emergent Adverse Events will be graded using the Common Terminology Criteria for Adverse Events (CTCAE) v. 5.0. Safety, tolerability, satisfaction, and quality of life assessed using the European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire 30 (EORTC QLQ-C30) questionnaire, as well as the PRO-CTCAE (Patient reported outcomes - Common Terminology Criteria for Adverse Events) questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Humaria Sarfraz, MD, Principal Investigator — The University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States